CLINICAL TRIAL: NCT06833216
Title: A Real-world Study of Familial Hereditary Breast Cancer in China
Brief Title: Familial Breast Cancer in China
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Head of department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5164
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Breast Carcinoma; Genetic Variation
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Familial breast cancer: Familial inherited breast cancer with genetic variants, including but not limited to mutations in the BRCA1, BRCA2, TP53, and PALB2 genes
  Interventions: Other: Genetic variation

INTERVENTIONS:
Other: Genetic variation — To observe and describe the clinical features, diagnosis and treatment plan and survival prognosis of familial hereditary breast cancer in China, and explore the main factors affecting prognosis.

SUMMARY:
This study is a retrospective descriptive study to collect clinical data (mainly including medical records and follow-up information, etc.) of breast cancer patients with genetic variation who were first diagnosed and treated in a number of hospitals in China during the period from January 1, 2015 to December 31, 2024, and to establish a retrospective cohort of familial hereditary breast cancer. To analyze the clinical features, diagnosis and treatment and survival prognosis of patients with familial hereditary breast cancer. To explore the main factors affecting clinical diagnosis and treatment and survival prognosis of patients

ELIGIBILITY:
Inclusion Criteria:

* Familial inherited breast cancer with genetic variants, including but not limited to mutations in the BRCA1, BRCA2, TP53, and PALB2 genes
* The patient had no major organ dysfunction
* ECOG score 0-1

Exclusion Criteria:

* There are serious dysfunction of vital organs (heart, liver, kidney)
* Patients with other malignancies, except cured non-melanoma skin cancer, cervical carcinoma in situ and other tumors that have been cured for at least 5 years
* In other acute infectious disease or chronic infectious disease activity period
* A history of uncontrolled seizures, central nervous system disorders, or mental disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 1, 2015 to December 31, 2024, a number of hospitals in China first diagnosed and treated breast cancer patients with genetic variants
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China